CLINICAL TRIAL: NCT02329080
Title: An International Phase II Trial Assessing Tolerability and Efficacy of Sequential Methotrexate-Aracytin-based Combination and R-ICE Combination, Followed by HD Chemotherapy Supported by ASCT, in Patients With Systemic B-cell Lymphoma With CNS Involvement at Diagnosis or Relapse (MARIETTA Regimen)
Brief Title: New Combination of Chemoimmunotherapy for Systemic B-cell Lymphoma With Central Nervous System Involvement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG42
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Methotrexate; Rituximab; Cytarabine; Thiotepa; Etoposide; Ifosfamide; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MATRIX - R-ICE - Conditioning and ASCT (Experimental): MATRIX (courses 1,2,3): Rituximab 375 mg/m2 d0/Methotrexate 3.5 g/m2 d1/Cytarabine 2 g/m2 d2 & d3/Thiotepa 30 mg/m2 d4/Liposomial Cytarabine 50 mg* d5
  R-ICE (courses 4,5,6):Rituximab 375 mg/m2 d1/Etoposide 100 mg/m2 d1,d2, d3/Ifosfamide 5 g/m2 d2/Carboplatin 5 AUC d2/Liposomial Cytarabine 50 mg* d4
  *If liposomal cytarabine is not available, standard intrathecal chemotherapy with methotrexate 10 mg + cytarabine 40 mg + hydrocortisone 50 mg can be administered. Oral steroids are suggested for 2-3 days after intrathecal liposomial cytarabine delivery to prevent chemical or aseptic meningitis/ arachnoiditis.
  Conditioning and ASCT: BCNU (carmustine)** 400 mg/m2 d-6/Thiotepa 5 mg/kg d-5 & d-4 ASCT: 5 x 106 CD34+cells/kg d0
  **In case of BCNU unavailability, the recommended conditioning regimen (Phase IV) is: Thiotepa 5 mg/kg d-6 & d-5/Busulfan 3.2 mg/kg d-4,d -3,d-2/Clonazepam 2 mg/d d-4,d -3,d-2 ASCT: 5 x 106 CD34+cells/kg d0
  Interventions: Drug: Methotrexate; Drug: Rituximab; Drug: Cytarabine; Drug: Thiotepa; Drug: liposomial cytarabine; Drug: Etoposide; Drug: Ifosfamide; Drug: Carmustine; Radiation: whole brain radiotherapy

INTERVENTIONS:
Drug: Methotrexate — methotrexate 3.5 g/m2 on day 1 courses 1, 2,3 of MATRIX regimen
Drug: Rituximab — Rituximab 375 mg/m2 as conventional IV infusion on day 0 courses 1, 2,3 (MATRIX regimen) and on day 1 courses 4,5,6 (R-ICE)
Drug: Cytarabine — Cytarabine 2 g/m2 every 12 hours, in 3-hr infusion on days 2,3 courses 1, 2,3 (MATRIX regimen)
Drug: Thiotepa — Thiotepa 30 mg/m2 in 30 minutes infusion on day 4 courses 1, 2,3 (MATRIX regimen) and 5 mg/kg in 250 ml of saline sol. in 2-hrs infusion every 12 hours on day -5 and -4 of conditioning and ASCT
Drug: liposomial cytarabine — Intrathecal liposomial cytarabine 50 mg on day 5 courses 1, 2,3 (MATRIX regimen) and on day 4 courses 4,5,6 (R-ICE)
Drug: Etoposide — Etoposide 100 mg/m2/d in 500 mL saline sol. in 30 minutes on day 1-2-3 courses 4,5,6 (R-ICE)
Drug: Ifosfamide — Ifosfamide 5 g/m2 in 1.000 mL saline sol. in 24-hour infusion on day 2 courses 4,5,6 (R-ICE)
Drug: Carmustine — BCNU (carmustine) 400 mg/m2 in 500 mL glucose 5% sol. in 1-hr infusion on day-6 of conditioning and ASCT
Radiation: whole brain radiotherapy — whole-brain irradiation 36 Gy + tumor- bed boost 10 Gy in patients with residual disease in the parenchymal brain/cerebellum.

SUMMARY:
This is an open, non comparative, multicentre phase II trial, to evaluate the efficacy and feasibility of a new sequential combination of HD-MTX-AraC-based chemoimmunotherapy, followed by R-ICE regimen, and by high-dose chemotherapy supported by ASCT.

DETAILED DESCRIPTION:
Treatment includes 6 courses of chemoimmunotherapy, the first three courses with an high dose methotrexate-based combination (MATRIX) followed by other three courses of R-ICE combination and finally a BCNU-thiotepa- containing conditioning and subsequent autologous stem cell transplantation.

MATRIX (courses 1, 2, 3):

Rituximab 375 mg/m2, Methotrexate 3.5 g/m2, Cytarabine 2 g/m2, Folinic rescue 15 mg/m2, Thiotepa 30 mg/m2, Intrathecal liposomial cytarabine 50 mg, rHuG-CSF 2,5 g/kg s.c.

R-ICE (courses 4, 5, 6):

Rituximab 375 mg/m2, Etoposide 100 mg/m2/d , Ifosfamide 5 g/m2, Intrathecal liposomial cytarabine 50 mg

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of diffuse large B-cell lymphoma
2. CNS involvement (brain, meninges, cranial nerves, eyes and/or spinal cord) at diagnosis (concomitant to extra-CNS disease) or relapse after conventional chemo(-immuno)therapy
3. Diagnosis of CNS involvement either by brain biopsy or CSF cytology examination. Neuroimaging alone is acceptable when stereotactic biopsy is formally contraindicated or when the disease has been previously histologically documented in other areas and the CNS localization is concomitant with a diffuse progression of systemic disease.
4. No previous treatment with high-dose methotrexate-based chemotherapy and/or brain irradiation. One-two courses of R-CHOP combination as upfront therapy are admitted in patients with large amount and/or extensive extra-CNS disease that could condition prognosis in an early phase of treatment. Local investigator decides if initial R-CHOP is needed based on patient's conditions
5. Age 18-70 years
6. ECOG performance status 0-3
7. Adequate bone marrow (Platelets count ≥100.000/mm3, hemoglobin ≥9 g/dL, neutrophils count≥1.500/mm3), renal (creatinine clearance ≥60 mL/min), cardiac (LVEF ≥50%), and hepatic function (total serum bilirubine ≤3 mg/dL, AST/ALT and GGT ≤2.5 per upper normal limit value), unless the abnormality is due to lymphoma infiltration
8. Absence of HIV infection and of detectable HCV-RNA and/or HBsAg and/or HBV-DNA
9. No concurrent malignancies. Previous malignancies are accepted if surgically cured or if there was no evidence of disease in the last 3 years at a regular follow-up
10. Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
11. Female patients must be non-pregnant and non-lactating. Sexually active patients of childbearing potential must implement adequate contraceptive measures during study participation
12. No treatment with other experimental drugs within the 6 weeks previous to enrolment
13. Given written informed consent prior to any study specific procedures, with the understanding that the patient has the right to withdraw from the study at any time, without any prejudice. Informed consent signed by a patient's guardian is acceptable if the patient is not able to decide inclusion in the study due to cognitive impairment

Exclusion Criteria:

1. Other lymphoma categories other than diffuse large B-cell lymphoma. In particular, patients with primary mediastinal lymphoma, intravascular large B-cell lymphoma or leg-type large B-cell lymphoma are excluded.
2. Patients with positive flow cytometry examination of the CSF, but negative results in CSF conventional cytology, and without any other evidence of CNS disease.
3. Patients with exclusive CNS disease at presentation (primary CNS lymphoma) are excluded
4. Previous treatment with support of autologous or allogeneic stem cells/bone marrow transplantation.
5. Symptomatic coronary artery disease, cardiac arrhythmias not well controlled with medication or myocardial infarction within the last 6 months (New York Heart Association Class III or IV heart disease)
6. Any other serious medical condition which could impair the ability of the patient to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-12; Primary Completion 2019-08 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrés JM Ferreri, MD, Study Chair — IELSG
Locations (36):
- Czechia (3):
  - Facultni nemocnice, Brno
  - FNKV (Facultni Nemocnice Kralovske Vinohrady), Prague
  - Vseobecna facultni nemocnice v Praze, Prague
- Italy (27):
  - Spedali Civili, Brescia
  - UO Ematologia e CTMO, PO Businco, Cagliari
  - IRST Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - UO Ematoliga Ospedale dell'Angelo, Mestre
  - San Raffaele H Scientific Institute, Milan
  - Istituto Nazionale Tumori, Milan
  - Ospedale Maggiore Policlinico, Milan
  - AOU Policlinico di Modena, Modena
  - SCDU Ematologia, Novara
  - Ematologia ed Immunologia Clinica - AO di Padova, Padua
  - UO Oncoematologia Ospedale Tortora, Pagani
  - Villa Sofia - Cervello, Palermo
  - Ematologia AOU, Parma
  - Ematologia Ospedale S.Maria delle Croci, Ravenna
  - A.O. Bianchi-Melacrino-Morelli, Divisione di Ematologia, Reggio Calabria
  - Arcispedale Santa Maria Nuova, Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Ematologia Università La Sapienza, Roma
  - IRCCS Istituto Regina Elena (IFO), Roma
  - Policlinico Universitario Campus Bio-Medico, Rome
  - IRCCS Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - AOU Senese, Siena
  - AO S.Maria di Terni, Terni
  - SC Ematologia AO Città della Salute e della Scienza, Torino
  - UO Ematologia Ospedale Panico, Tricase
  - AOU Santa Maria della Misericordia, Udine
  - UOC Ematologia Policlinico Rossi, Verona
  - Ematologia Ospedale S. Bortolo, Vicenza
- Erasmus MC, Rotterdam, Netherlands
- United Kingdom (5):
  - Beatson Cancer Center, Glasgow
  - Liverpool Aintree, Liverpool
  - UCLH University College London Hospitals NHS foundation trust, London
  - The Christie Hospital, Manchester
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Ferreri AJM, Doorduijn JK, Re A, Cabras MG, Smith J, Ilariucci F, Luppi M, Calimeri T, Cattaneo C, Khwaja J, Botto B, Cellini C, Nassi L, Linton K, McKay P, Olivieri J, Patti C, Re F, Fanni A, Singh V, Bromberg JEC, Cozens K, Gastaldi E, Bernardi M, Cascavilla N, Davies A, Fox CP, Frezzato M, Osborne W, Liberati AM, Novak U, Zambello R, Zucca E, Cwynarski K; International Extranodal Lymphoma Study Group (IELSG). MATRix-RICE therapy and autologous haematopoietic stem-cell transplantation in diffuse large B-cell lymphoma with secondary CNS involvement (MARIETTA): an international, single-arm, phase 2 trial. Lancet Haematol. 2021 Feb;8(2):e110-e121. doi: 10.1016/S2352-3026(20)30366-5. PMID 33513372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the recruitment period 79 patients were enrolled and 75 of them were treated.
  Four patients were excluded after enrolment before the start of study treatment because of unrelated laboratory abnormalities (two patients), disease only at flow cytometry examination of the cerebrospinal fluid (one), and death at the same time as registration (one).
Period: Overall Study
Arm/Group | MATRIX - R-ICE - Conditioning and ASCT
Started | 75
Completed | 37
Not Completed | 38
Not completed — Adverse Event | 1
Not completed — Death | 4
Not completed — Lack of Efficacy | 22
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Partial response | 4
Not completed — Complete response | 4

BASELINE CHARACTERISTICS:
Arm/Group | MATRIX - R-ICE - Conditioning and ASCT
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 4
  Italy | 52
  United Kingdom | 18
  Switzerland | 1
CNS involvement at presentation [Count of Participants; unit: Participants]
  CNS involvement at presentation | 32
  No CNS involvement at presentation | 43
Isolated CNS relapse [Count of Participants; unit: Participants]
  Isolated CNS relapse | 15
  No isolated CNS relapse | 60
Concomitant CNS-systemic localisation [Count of Participants; unit: Participants]
  Concomitant CNS-systemic localisation | 28
  No concomitant CNS-systemic localisation | 47
HBV or HCV seropositivity [Count of Participants; unit: Participants]
  HBV or HCV seropositivity | 2
  No HBV or HCV seropositivity | 73
CNS site of disease - Brain parenchima [Count of Participants; unit: Participants]
  Brain parenchima | 34
  No brain parenchima | 41
CNS site of disease - Cerebrospinal fluid or meninges [Count of Participants; unit: Participants]
  Cerebrospinal fluid or meninges | 8
  No cerebrospinal fluid or meninges | 67
CNS sites of disease - Spinal cord [Count of Participants; unit: Participants]
  Spinal cord | 2
  No spinal cord | 73
CNS sites of disease - Eyes [Count of Participants; unit: Participants]
  Eyes | 2
  No eyes | 73
CNS sites of disease - Brain and cerebrospinal fluid or meninges [Count of Participants; unit: Participants]
  Brain and cerebrospinal fluid or meninges | 13
  No brain and cerebrospinal fluid or meninges | 62
CNS sites of disease - Brain and eyes [Count of Participants; unit: Participants]
  Brain and eyes | 10
  No Brain and eyes | 65
CNS sites of disease - Brain, cerebrospinal fluid and eyes [Count of Participants; unit: Participants]
  Brain, cerebrospinal fluid and eyes | 6
  No brain, cerebrospinal fluid and eyes | 69
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) [Count of Participants; unit: Participants] — Patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability graded as follows:
  0: Fully active, able to carry on all pre-disease performance without restriction;
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature;
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities;
  3. Capable of only limited selfcare;
  4. Completely disabled; totally confined to bed or chair;
  5. Dead
  Participants
    ECOG-PS > 1 | 28
    ECOG-PS </= 1 | 47
Number of extranodal organs involved (other than CNS) [Count of Participants; unit: Participants]
  Number of extranodal organs involved >1 | 23
  Number of extranodal organs involved </=1 | 52
High LDH serum concentration [Count of Participants; unit: Participants]
  High LDH serum concentration | 37
  No high LDH serum concentration | 38
Advanced stage [Count of Participants; unit: Participants]
  Advanced stage | 60
  No advanced stage | 15
International Prognostic Index (IPI) [Count of Participants; unit: Participants]
  Low IPI risk | 14
  Low-intermediate IPI risk | 18
  High-intermediate IPI risk | 26
  High IPI risk | 17

OUTCOME MEASURES:

1. Primary Outcome: 1 Year Progression Free Survival (PFS)
Description: Percentage of patients free from progression after 1 year from study entry
Time Frame: From study entry until 1 year after
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MATRIX - R-ICE - Conditioning and ASCT
Number analyzed (Participants) | 75
Percentage of participants | 58 [55 to 61]

2. Secondary Outcome: 2 Years Progression Free Survival (PFS)
Description: Percentage of patients free from progression after 2 years from study entry
Time Frame: From study entry until 2 years after
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MATRIX - R-ICE - Conditioning and ASCT
Number analyzed (Participants) | 75
percentage of participants | 46 [39 to 53]

3. Secondary Outcome: 2 Years Overall Survival (OS)
Description: Percentage of participants alive after 2 years from study entry
Time Frame: From trial entry until 2 years after
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MATRIX - R-ICE - Conditioning and ASCT
Number analyzed (Participants) | 75
percentage of participants | 46 [39 to 53]

ADVERSE EVENTS:
Time Frame: All cause mortality was assessed through 2 years after study entry. All AEs were collected from trial inclusion until 30 days after end of treatment (7 months)
Groups:
- Enrolled, But Not Treated: Four patients were excluded after enrolment
Arm/Group | MATRIX - R-ICE - Conditioning and ASCT | Enrolled, But Not Treated
All-Cause Mortality (participants affected / at risk) | 50/75 | 1/4
Serious Adverse Events (participants affected / at risk) | 46/75 | 0/4
Other Adverse Events (participants affected / at risk) | 72/75 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MATRIX - R-ICE - Conditioning and ASCT (N=75) | Enrolled, But Not Treated (N=4)
Alanine aminotransferase increased (Investigations) | 1 (1) | NA
Hyponatremia (Investigations) | 1 (1) | NA
Poorly differentiated adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA
Bleeding (Vascular disorders) | 1 (1) | NA
Thromboembolic event (Vascular disorders) | 1 (1) | NA
Deep vein thrombosis (Vascular disorders) | 1 (1) | NA
Atrial fibrillation (Cardiac disorders) | 1 (1) | NA
Neurological toxicity (Nervous system disorders) | 1 (1) | NA
Brain ischemic stroke (Nervous system disorders) | 1 (1) | NA
Encephalopathy (Nervous system disorders) | 1 (1) | NA
Bleeding brain lesion (Nervous system disorders) | 1 (1) | NA
Fatigue (General disorders) | 1 (1) | NA
Fever (General disorders) | 1 (2) | NA
Pain (General disorders) | 1 (1) | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (23) | NA
Neutropenic fever (Blood and lymphatic system disorders) | 3 (4) | NA
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | NA
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | NA
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2) | NA
Vomiting and diarrhea (Gastrointestinal disorders) | 1 (2) | NA
Microperforation of the bowel (Gastrointestinal disorders) | 1 (1) | NA
Bowel perforation (Gastrointestinal disorders) | 1 (1) | NA
Acute renal failure (Renal and urinary disorders) | 1 (1) | NA
Acute kidney injury (Renal and urinary disorders) | 1 (1) | NA
Septic arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | NA
Septic shock (Infections and infestations) | 3 (3) | NA
Interstitial pneumonia (Infections and infestations) | 1 (1) | NA
Sepsis (Infections and infestations) | 13 (15) | NA
Pneumonia (Infections and infestations) | 3 (3) | NA
Cytomegalovirus infection (Infections and infestations) | 1 (1) | NA
Cytomegalovirus reactivation (Infections and infestations) | 1 (2) | NA
Neutropenic sepsis (Infections and infestations) | 2 (2) | NA
Adenovirus infection (Infections and infestations) | 1 (1) | NA
Fungal chest infection (Infections and infestations) | 1 (1) | NA
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | NA
Catheter related infection (Infections and infestations) | 1 (1) | NA
Tuberculosis (Infections and infestations) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MATRIX - R-ICE - Conditioning and ASCT (N=75) | Enrolled, But Not Treated (N=4)
Vascular Disorders (Vascular disorders) | 15 (23) | NA
Cardiac Disorders (Cardiac disorders) | 8 (16) | NA
Nervous System Disorders (Nervous system disorders) | 24 (67) | NA
Blood and Lymphatic System Disorders G3-4 (Blood and lymphatic system disorders) | 51 (327) | NA
General Disorders and Administration Site Conditions (General disorders) | 55 (121) | NA
Eye Disorders (Eye disorders) | 5 (6) | NA
Gastrointestinal Disorders (Gastrointestinal disorders) | 35 (116) | NA
Respiratory Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 9 (13) | NA
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 15 (15) | NA
Renal and Urinary Disorders (Renal and urinary disorders) | 7 (12) | NA
Infections and Infestations (Infections and infestations) | 28 (65) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02329080/Prot_SAP_000.pdf